CLINICAL TRIAL: NCT01352377
Title: A STUDY ASSESSING THE IMPACT OF THE NEW CLSI GUIDELINES ON ANTIBIOTIC SUSCEPTABILITY TESTING PATTERNS
Brief Title: Impact of New CLSI Guidelines on Antibiotic Susceptability Pattern
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Southern Nevada (Other)
Responsible Party: Alan Greenberg, UMC
Other Study IDs: P20RR016464 (NIH)
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-04

CONDITIONS: Antibiotic Susceptibility Patterns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Assessing the precise MIC for the Ceftriaxone using E-test. To determine what proportion of susceptibility reports will be reclassified based on the new CLSI guidelines.Antibiotic susceptibility reports of blood cultures, urine cultures,aseptic body fluid cultures growing Enterobacteriaceae organism generated by the Phoenix machine will be obtained on a daily basis.MIC for Ceftriaxone will be noted.If the MIC is <=2 for Ceftriaxone,those cultures would be used to run an additional test - E- test.E-test gives us more precise MIC values compared to Phoenix machine.We will analyze the data collected over 2 months. We will determine the proportion of susceptibility reports reclassified based on the new CLSI guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Antibiotic susceptibility reports of blood cultures, urine cultures,aseptic body fluid cultures growing Enterobacteriaceae organism generated by the Phoenix machine.

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age more than 21 years who are inpatients at UMC.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Umc, Las Vegas, Nevada, United States